CLINICAL TRIAL: NCT06007417
Title: The Efficacy and Safety of Once-weekly PEG-somatropin (GenSci004) in Treatment-naive Children With Growth Hormone Deficiency: A Randomized, Open-label, Parallel-group, Active-Controlled, Non-inferiority Phase 3 Study (ELEVATE)
Brief Title: A Study to Investigate Efficacy and Safety of Weekly PEG-somatropin (GenSci004) in Treatment Naive Children With Growth Hormone Deficiency
Acronym: ELEVATE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GenSci004-301
Record Dates: First submitted 2023-08-09; First posted 2023-08-23 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: GHD
Keywords: GHD; growth hormone deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- GenSci004 (Experimental)
  Interventions: Drug: GenSci004
- Genotropin (Active Comparator)
  Interventions: Drug: Genotropin

INTERVENTIONS:
Drug: GenSci004 — GenSci004 is a pegylated rhGH (PEG rhGH) (i.e., PEG-somatropin)
  Arms: GenSci004
Drug: Genotropin — Genotropin
  Arms: Genotropin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of weekly GenSci004 compared with daily Genotropin in treatment-naive children with growth failure due to GHD.

DETAILED DESCRIPTION:
The purpose of this Phase 3 study is to evaluate the efficacy, safety, and tolerability of weekly GenSci004 compared to daily Genotropin over 52 weeks in prepubertal treatment-naïve children with growth failure due to GHD.

ELIGIBILITY:
Inclusion Criteria:

1. Prepubertal children with GHD in Tanner Stage 1
2. Baseline HT at least -2.0 SD below the mean HT for CA and sex (HT SDS ≤ 2.0).
3. Body mass index (BMI) within ±2.0 SD of the mean BMI for BA and sex.
4. Growth hormone stimulation tests: ≤10 ng/mL
5. Baseline IGF 1 level of at least 1.0 SD below the mean IGF 1 level standardized for age and sex (IGF 1 SDS ≤-1.0)
6. Normal 46 XX karyotype for girls.
7. Children with multiple hormonal deficiencies must be on stable replacement therapy for other hypothalamo-pituitary axes for at least 3 months
8. Written, signed informed consent of the parent(s) or legal guardian(s) of the participant and written assent of the participant

Exclusion Criteria:

1. BA≥CA
2. Prior exposure to rhGH, long-acting growth hormones, or IGF 1 therapy.
3. Major medical conditions or presence of contraindication to human growth hormone (hGH) treatment
4. Participation in any other trial of an investigational agent within 3 months prior to Screening.
5. Any reason per investigator's discretion

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 162 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Annualized Height Velocity (AHV) for GenSci004 and Genotropin groups | 52 weeks
  Measured in centimeter per year (cm/year)

SECONDARY OUTCOMES:
Annualized Height Velocity (AHV) for GenSci004 and Genotropin groups | 104 weeks
  Measured in centimeter per year (cm/year)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Miller, Study Chair — University of Minnesota
Locations (1):
- Cook Childrens, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No